CLINICAL TRIAL: NCT02982213
Title: Presence of a Companion During Performance of Neuraxial Labor Analgesia
Acronym: Companion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Feyce M. Peralta, MD, MS, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00203896
Record Dates: First submitted 2016-11-16; First posted 2016-12-05 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Anxiety; Pain; Health Knowledge, Attitudes, Practice
Keywords: Newest Vital Sign; Anxiety; Health literacy; Neuraxial Analgesia; Epidural catheter placement; Pregnancy; Parturients; Pain Catastrophizing Scale; STAI questionnaire; Companion
MeSH Terms: conditions — Anxiety Disorders; Pain; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No companion present (No Intervention): No companion is present during the placement of the epidural catheter.
- Companion present (Active Comparator): A companion will be present during the placement of the epidural catheter.
  Interventions: Other: Companion Present

INTERVENTIONS:
Other: Companion Present — A companion will be present during the epidural catheter placement.
  Arms: Companion present

SUMMARY:
The purpose of the study is to evaluate if maternal anxiety is improved when a parturient gets her choice with regard to the presence of a companion during epidural catheter placement for labor analgesia. It will be focused on parturients having their first child with the current partner. Additionally, it will investigate the effect of ethnicity, health literacy (as evaluated by the Newest Vital Sign questionnaire), catastrophizing (as evaluated by the Pain Catastrophizing Scale), and the relationship of the support person to the parturient. The investigators hypothesize that there may be specific subgroups in which maternal anxiety is improved when a parturient gets her choice regarding the presence of a companion during labor epidural catheter placement; however, a significant improvement in maternal anxiety, when including all participants, will not be appreciated.

DETAILED DESCRIPTION:
Parturients who have been admitted to the Labor and Delivery ward at Prentice Women's Hospital will be approached by a member of the anesthesia team prior to the placement of a labor epidural catheter. They will be asked if they are considering neuraxial labor analgesia, and if they are they will be screened using the inclusion and exclusion criteria to determine study eligibility. Once they have been evaluated and found to be appropriate for the study, they will be invited to participate.

Participants will be asked to fill out the STAI questionnaire to assess the level of anxiety prior to placement of the labor epidural catheter, and before knowing their group assignment. They will then complete the pre procedure questionnaire. This questionnaire asks about expectations she has for the labor epidural procedure. They will then be given the page of the Newest Vital Signs questionnaire with the Nutrition Facts, and be asked the 6 questions by the recruiter. Then they will be handed the Pain Catastrophizing Scale form with 13 statements, and asked to fill it out as directed in the instructions at the top. They will then be asked who their primary support person is. A form will be handed to that person to confidentially record if he/she would prefer to be present for the procedure. This form will be collected from the companion, and without the parturient aware of the support person's response, she will be asked for her preference with regard to the presence of a companion in the room, which will be recorded on this form as well. Finally, she will be asked which ethnicity she most relates to, also to be recorded on this form.

After all these data have been collected, the parturient will be randomized as to whether her companion will be allowed in the room or will be asked to leave. This will not be communicated to the parturient until the time of the labor epidural catheter placement. When she requests the neuraxial labor analgesia, the provider placing the labor epidural catheter will be made aware of which group she has been randomized to, and will either ask the companion to leave for placement, or provide the support person a non-mobile chair to sit on in front of the parturient for placement of the labor epidural. The companion will be asked to remain in the chair. He/she will be asked to focus on the parturient. It will be emphasized that he/she must remain seated and will not be allowed to observe the procedure being performed. This is to prevent loss of consciousness in the support person, which has been documented in the literature (Devore and Asrani, 1978; Crosby and Halpern, 1989). One violation will result in a warning, and after a second the companion will be escorted out of the room and the participant will be removed from the study.

The provider will place the labor epidural catheter in the regular fashion, as is common practice at Prentice Women's Hospital. After preparation and draping of the skin in the sitting position, infiltration with Lidocaine 1% will be conducted at L3-L4 or L4-L5. A 17g Tuohy needle will be advanced into the epidural space, using a loss of resistance with either saline or air, depending on the provider's preference. After the epidural space has been located, a 27g pencil-tip spinal needle will be placed through the Tuohy, into the intrathecal space, and an intrathecal dose of medication will be administered. The exact dose to be injected will be left up to the discretion of the provider, who will determine the appropriate dose based on the patient's situation at that time. After the intrathecal dose is administered, the spinal needle will be removed and a 19g epidural catheter will be placed through the Tuohy into the epidural space. It will be secured at the skin with a sterile dressing and tape, leaving 5cm of the catheter in the epidural space. The patient will then be placed in a lateral position.

After the completion of the neuraxial procedure, the study participant will then be asked to fill out the STAI questionnaire again. Additionally, she will be asked to record her perception of pain during the placement of the labor epidural catheter, using a VAS (Visual Analogue Scale) from 0-100mm. At that point the parturient's participation in the study will be complete.

The provider placing the labor epidural catheter will be asked to evaluate his/her ability to palpate landmarks for placement, the positioning of the patient, and overall perceived difficulty with the epidural placement, using a VAS from 0-100mm for each, which will be kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* Delivering the first child
* Planning to labor with neuraxial analgesia.
* Additionally, there will need to be sufficient time before delivery to allow the completion of the Pre procedure questionnaire, State-Trait Anxiety Inventory (STAI) questionnaire both before and after the procedure, as well as the Newest Vital Sign questionnaire and the Pain Catastrophizing Scale questionnaire before the procedure.
* They will be included if they are ASA (American Society of Anesthesiologists) 2.
* Able to read and comprehend the English language, as the Newest Vital Sign questionnaire requires them to read and interpret a nutrition label.

Physician Inclusion:

* Anesthesiology Attending Physician, fellow or resident who participants in the placement of the epidural catheter placement

Companion Inclusion:

* Primary companion identified by parturient over the age of 18

Exclusion Criteria:

* Parturients will be excluded if they are receiving neuraxial anesthesia for a cesarean delivery,
* External cephalic version
* Non-labor procedure.
* Subjects will be excluded if they begin to push for delivery before completion of the STAI questionnaire following labor epidural catheter placement.
* They will be excluded if there is no support person present at the time of the neuraxial procedure.
* They will be excluded if they are ASA 3 or greater, or if they have a contraindication to receiving any of the medications routinely used in the placement of a labor epidural catheter (lidocaine, bupivacaine, epinephrine, fentanyl).
* Adults who are unable to consent and minors will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feyce Peralta, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Companion Present | Companion Present
Started | 75 | 75
Completed | 70 | 74
Not Completed | 5 | 1
Not completed — Did not complete follow up questionnaire | 5 | 1

BASELINE CHARACTERISTICS:
Population: In the companion not in the room group, 73 subjects received the intervention and 70 completed follow up.
  In the companion in the room group, 75 completed demographic data, 73 subjects received intervention and 74 completed follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Companion Present | Companion Present | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: In the companion not in the room group, 73 completed demographic data, 73 subjects received the intervention and 70 completed follow up.In the companion in the room group, 75 completed demographic data, 75 subjects received intervention and 74 completed follow up.
  years
    number analyzed (Participants) | 73 | 75 | 148
    (all) | 32.2 (3.8) | 31.8 (3.6) | 32 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 52 | 48 | 100
  African American | 4 | 5 | 9
  Asian | 11 | 11 | 22
  Latino/Hispanic | 6 | 10 | 16
  Question not answered | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 147
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.2 (4.7) | 29.6 (7.3) | 29.4 (6.1)
Gestational Age [Mean (Full Range); unit: Weeks] — Population: In the companion not in the room group 72 completed gestational data and in the companion group 73 completed the gestational data. .
  Weeks
    number analyzed (Participants) | 72 | 73 | 145
    (all) | 40 [39 to 41] | 40 [39 to 41] | 40 [39 to 41]
NRS pain score [Mean (Full Range); unit: units on a scale] — Numerical Rating Scale (NRS) pain score (0 no pain to 10 worst pain imaginable) at request for neuraxial analgesia Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery
  units on a scale
    number analyzed (Participants) | 73 | 74 | 147
    (all) | 7 [6 to 8] | 7 [6 to 8] | 7 [6 to 8]
Cervical Dilation [Mean (Full Range); unit: centimeters] — Cervical dilation in centimeters. Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed .
  centimeters
    number analyzed (Participants) | 73 | 74 | 147
    (all) | 3 [2 to 4] | 3.5 [2 to 4.5] | 3 [2 to 4.5]
Labor Type [Count of Participants; unit: Participants] — Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery)
  Participants
    Induction: number analyzed (Participants) | 73 | 74 | 147
    Induction | 44 | 38 | 82
    Spontaneous labor: number analyzed (Participants) | 73 | 74 | 147
    Spontaneous labor | 29 | 36 | 65
Labor epidural procedural expectations [Count of Participants; unit: Participants] — Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery)
  Participants
    None: number analyzed (Participants) | 73 | 74 | 147
    None | 4 | 4 | 8
    Short procedure minimal pain: number analyzed (Participants) | 73 | 74 | 147
    Short procedure minimal pain | 49 | 53 | 102
    Long procedure pain not mentioned: number analyzed (Participants) | 73 | 74 | 147
    Long procedure pain not mentioned | 3 | 0 | 3
    Painful procedure: number analyzed (Participants) | 73 | 74 | 147
    Painful procedure | 13 | 13 | 26
    Other than pain or duration: number analyzed (Participants) | 73 | 74 | 147
    Other than pain or duration | 4 | 4 | 8
Greatest concern regarding epidural procedure [Count of Participants; unit: Participants] — Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section).
  Participants
    Pain during procedure: number analyzed (Participants) | 73 | 75 | 148
    Pain during procedure | 23 | 20 | 43
    Unable to tolerate procedure: number analyzed (Participants) | 73 | 75 | 148
    Unable to tolerate procedure | 4 | 4 | 8
    Ineffective analgesia: number analyzed (Participants) | 73 | 75 | 148
    Ineffective analgesia | 17 | 14 | 31
    Complications: number analyzed (Participants) | 73 | 75 | 148
    Complications | 23 | 28 | 51
    Other: number analyzed (Participants) | 73 | 75 | 148
    Other | 6 | 9 | 15
Have you spoken to friends or family about labor epidurals? [Count of Participants; unit: Participants] — Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery)
  Participants
    Yes-positive comments: number analyzed (Participants) | 73 | 74 | 147
    Yes-positive comments | 53 | 49 | 102
    Yes-mixed comments: number analyzed (Participants) | 73 | 74 | 147
    Yes-mixed comments | 13 | 13 | 26
    Yes-mostly negative comments: number analyzed (Participants) | 73 | 74 | 147
    Yes-mostly negative comments | 1 | 3 | 4
    Did not respond: number analyzed (Participants) | 73 | 74 | 147
    Did not respond | 6 | 9 | 15
Researched epidurals through social media? [Count of Participants; unit: Participants] — Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery)
  Participants
    Yes: number analyzed (Participants) | 73 | 74 | 147
    Yes | 37 | 43 | 80
    No: number analyzed (Participants) | 73 | 74 | 147
    No | 36 | 31 | 67
Relationship of primary companion [Count of Participants; unit: Participants]
  Male partner | 62 | 65 | 127
  Female partner | 10 | 6 | 16
  Brother | 1 | 0 | 1
  Aunt | 0 | 1 | 1
  Friend | 2 | 3 | 5
How long have you known your companion (years)? [Mean (Full Range); unit: Years] — Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery)
  Years
    number analyzed (Participants) | 73 | 74 | 147
    (all) | 7.5 [6 to 11] | 7 [5 to 11] | 7 [5 to 11]
Work in medical field? [Count of Participants; unit: Participants] — Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery)
  Participants
    Yes: number analyzed (Participants) | 73 | 74 | 147
    Yes | 12 | 12 | 24
    No: number analyzed (Participants) | 73 | 74 | 147
    No | 61 | 62 | 123
Preprocedure pain catastrophizing scale [Median (Inter-Quartile Range); unit: units on a scale] — The PCS is a self reported 13 item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). The PCS is contains three subscales being magnification, rumination, and helplessness. Possible score is 0-52 where the higher scores indicate that the more catastrophizing thoughts are present. Catastrophizing thinking can result in a more intense experience of pain. Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery)
  units on a scale
    Median (quartile): number analyzed (Participants) | 73 | 74 | 147
    Median (quartile) | 12 [8 to 22] | 17 [11 to 22] | 14 [8 to 22]
    Upper (quartile): number analyzed (Participants) | 73 | 74 | 147
    Upper (quartile) | 18 [18 to 25] | 23 [23 to 31] | 21 [18 to 31]
Newest vital sign [Count of Participants; unit: Participants] — The Newest Vital Sign (NVS), is a nutrition label is accompanied by 6 questions. Answering more than 4 correct responses are unlikely to have low literacy, whereas answering fewer than 4 correct answers indicate the possibility of limited literacy. Possible score 0 low health literacy-6 high health literacy. Population: 74 in the partner in the room group were analysed (1 emergency cesarean delivery).
  Participants
    number analyzed (Participants) | 75 | 74 | 149
    Good health literacy | 62 | 65 | 127
    Low health literacy | 13 | 9 | 22
State-Trait (STAI) Anxiety Inventory [Mean (Full Range); unit: Score on a scale] — The State-Trait Anxiety Inventory (STAI) is used to measure of trait and state anxiety. There are 20 items for assessing trait anxiety and 20 for state anxiety. Both tests are scored on a 4-point scale (from "Almost Never" to "Almost Always"). Score limit for each test is 20 low to 80 high. Low to mild anxiety is a score of 20-37, moderate anxiety is a score of 38-44 and high anxiety is a score of 45-80. Population: 73 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery)
  Score on a scale
    State: number analyzed (Participants) | 73 | 74 | 147
    State | 38 [31 to 46] | 38 [32 to 50] | 38 [31 to 50]
    Trait: number analyzed (Participants) | 73 | 74 | 147
    Trait | 29 [26 to 35] | 31 [26 to 37] | 30 [26 to 37]
Labor Epidural Performance: Trainee Level [Count of Participants; unit: Participants] — Physician training level of the operator of the epidural placement catheter. Population: Training level of operator for the epidural catheter placement CA1-CA3 = clinical anesthesiology training year.
  70 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section 3 no follow up)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery).
  Participants
    Clinical Anesthesia 1: number analyzed (Participants) | 70 | 74 | 144
    Clinical Anesthesia 1 | 6 | 6 | 12
    Clinical Anesthesia 2: number analyzed (Participants) | 70 | 74 | 144
    Clinical Anesthesia 2 | 48 | 46 | 94
    Clinical Anesthesia 3: number analyzed (Participants) | 70 | 74 | 144
    Clinical Anesthesia 3 | 16 | 20 | 36
    Fellow: number analyzed (Participants) | 70 | 74 | 144
    Fellow | 0 | 2 | 2
Number of Participants Categorized by Number of Epidural Catheter Attempts [Count of Participants; unit: Participants] — Population: 70 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section 3 no follow up)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery).
  Participants
    1 Attempt: number analyzed (Participants) | 70 | 74 | 144
    1 Attempt | 59 | 65 | 124
    2 Attempts: number analyzed (Participants) | 70 | 74 | 144
    2 Attempts | 5 | 5 | 10
    Attempts not recorded: number analyzed (Participants) | 70 | 74 | 144
    Attempts not recorded | 6 | 4 | 10
Number of Attending Anesthesiologist Takeover of Epidural Placement [Number; unit: Attending Takeovers] — Population: 70 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section 3 no follow up)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery).
  Attending Takeovers
    number analyzed (Participants) | 70 | 74 | 144
    (all) | 8 | 4 | 12
Resident Assessment of Difficulty of Epidural Procedure [Median (Inter-Quartile Range); unit: Score on a scale] — Difficulty of procedure scored on a scale of 0 (extremely difficult) to 100 (not difficult). Population: 70 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section 3 no follow up)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery).
  Score on a scale
    number analyzed (Participants) | 70 | 74 | 144
    (all) | 80 [50 to 90] | 78 [44 to 90] | 79 [44 to 90]
Resident Assessment of Ability to Position Patient (0-100) [Median (Inter-Quartile Range); unit: units on a scale] — The operator (resident) assessment of the difficulty of preparing the patient for positioning prior to the epidural catheter placement scored on a scale of 0 (difficult) to 100 (easy). Population: 70 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section and 3 no follow up) and 74 in the partner in the room group were analysed (1 emergency cesarean delivery).
  units on a scale
    number analyzed (Participants) | 70 | 74 | 144
    (all) | 77 [65 to 90] | 78 [70 to 90] | 77 [65 to 90]
Resident Assessment of Ability to Palpate Landmarks [Median (Inter-Quartile Range); unit: units on a scale] — Operator (resident) assessment of ability to palpate landmarks prior to epidural placement procedure on a scale of 0 extremely difficult to 100 not difficult. Population: 70 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section and 3 no follow up)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery).
  units on a scale
    number analyzed (Participants) | 70 | 74 | 144
    (all) | 78 [50 to 93] | 70 [48 to 87] | 75 [48 to 93]
Resident Comfort Performing Procedure (0-10) [Median (Inter-Quartile Range); unit: units on a scale] — Operator (resident) comfort performing the epidural placement procedure on a scale of 0 (severe discomfort) to 10 being (extremely comfortable). Population: 70 in the no companion in the room were analysed (1 wd consent and 1 emergency c-section and 3 no follow up)and 74 in the partner in the room group were analysed (1 emergency cesarean delivery).
  units on a scale
    number analyzed (Participants) | 70 | 74 | 144
    (all) | 8 [6.5 to 9] | 8 [7 to 9] | 8 [6.5 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Maternal Satisfaction and the Presence of a Companion During the Placement of Epidural Catheter for Labor Analgesia.
Description: The maternal satisfaction after epidural catheter placement for labor analgesia and the presence of a companion scored on a 5 point Likert scale of Highly Dissatisfied, Dissatisfied, Neutral, Satisfied and Highly Satisfied
Time Frame: Average 12 hours, up to 24 hours after epidural placement
Measure: Count of Participants; unit: Participants
Arm/Group | No Companion Present | Companion Present
Number analyzed (Participants) | 70 | 74
Participants
  Highly Dissatisfied | 2 | 2
  Dissatisfied | 3 | 0
  Neutral | 11 | 1
  Satisfied | 15 | 10
  Highly Satisfied | 39 | 61
Statistical Analysis 1: Comparison: No Companion Present vs Companion Present; Test type: Superiority; p = .001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = .025

2. Secondary Outcome: Does the Desire of Subject to Have the Companion Present Affect the Anxiety of the Subject Measured Using the STAI (State-Trait Anxiety Inventory) Questionnaire.
Description: Analysis of maternal anxiety, pre and post placement of the epidural catheter, using the STAI questionnaire.The STAI is a two part 20 question per part anxiety scale survey. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. The State-Trait Anxiety Inventory (STAI) is used to measure of trait and state anxiety. There are 20 items for assessing trait anxiety and 20 for state anxiety. Both tests are scored on a 4-point scale (from "Almost Never" to "Almost Always"). Score limit for each test is 20 low to 80 high. Low to mild anxiety is a score of 20-37, moderate anxiety is a score of 38-44 and high anxiety is a score of 45-80. The score represents the difference between the pre STAI and the post procedure STAI in each group.
Time Frame: 24 hours after epidural placement
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | No Companion Present | Companion Present
Number analyzed (Participants) | 70 | 74
score on scale | -7 [-13 to -1] | -11 [-17 to -3]

3. Secondary Outcome: Does the Presence of a Companion Affect the Perceived Difficulty of the Procedure by the Resident Physician Placing the Labor Epidural Catheter.
Description: Analysis of the perceived difficulty for the anesthesia resident physician, through utilization of a scale of 0 (severe discomfort to 10 (extremely comfortable).
Time Frame: After epidural placement
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | No Companion Present | Companion Present
Number analyzed (Participants) | 70 | 74
score on scale | 8 [6.5 to 9] | 8 [7 to 9]

4. Secondary Outcome: What is the Preference of Subjects to Have a Companion Present for Future Procedures.
Description: What is the preference of subjects having a companion present using 5 point Likert like scale of highly unlikely to highly likely.
Time Frame: 24 hours after epidural placement
Measure: Count of Participants; unit: Participants
Arm/Group | No Companion Present | Companion Present
Number analyzed (Participants) | 73 | 74
Participants
  Highly likely | 17 | 30
  Likely | 14 | 15
  Neutral | 22 | 14
  Unlikely | 7 | 5
  Highly unlikely | 10 | 10
  Did not respond | 3 | 0

5. Secondary Outcome: Recommend Care Received Based on Experience of Companion Presence in Room During Epidural Procedure.
Description: Recommend care based on presence or absence of a companion received based on Likert type scale of highly unlikely to highly likely.
Time Frame: 24 hours after epidural
Measure: Count of Participants; unit: Participants
Arm/Group | No Companion Present | Companion Present
Number analyzed (Participants) | 73 | 74
Participants
  Highly likely | 32 | 59
  LIkely | 10 | 11
  Neutral | 22 | 2
  Unlikely | 3 | 0
  Highly unlikely | 3 | 2
  Did not respond | 3 | 0
Statistical Analysis 1: Comparison: No Companion Present vs Companion Present; Test type: Equivalence — Sample size of 5 per group to achieve 80% power to detect a change in the log odds ration of 1.0 at a .05 significance level using a two sided Mann Whitney U test; p = .001, McNemar

ADVERSE EVENTS:
Time Frame: 24 hours after delivery of the baby.
Description: Emotional distress answering some of the questionnaires as reported by the subject to the study team members.
Groups:
- No Companion: No companion in the room during the procedure
- Companion Present: Companion present during the procedure
Arm/Group | No Companion | Companion Present
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

LIMITATIONS AND CAVEATS:
The limitation is our sample was primarily Caucasian with mid to high socioeconomic status. Additionally, most of the companions were married to the study participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT02982213/Prot_SAP_000.pdf